CLINICAL TRIAL: NCT05335213
Title: Urinary Tract Infections in Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gomel State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2.15
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Liver Cirrhosis; Urinary Tract Infections
MeSH Terms: conditions — Liver Cirrhosis; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — The urine and fecal specimens collect and store at -80°C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with cirrhosis and urinary tract infections: Participants collect urine and fecal specimens at first two days when they admit to hospital, after 7-10 days and last two days hospital treatment and during episodes of complications (variceal bleeding, hepatic coma, hepatorenal syndrome).
  Urine samples take from patients via clean catch if the patient not have a catheter placed, otherwise take from urinary catheters if present. Straight catheterization utilize if the patient unable to void and doesn't have a catheter placed.
  Fecal specimens collect using a toilet specimen collection kit. Clinical, standart laboratory and cultural test, molecular genetic methods, using 16S rRNA gene sequencing of the V4-V5 hypervariable region be administered.
  Interventions: Diagnostic Test: 16S rRNA gene sequencing
- Participants with cirrhosis without urinary tract infections: Participants ask to collect urine and fecal specimens at first two days when they admit to hospital, after 7-10 days and last two days hospital treatment and during episodes of complications (variceal bleeding, hepatic coma, hepatorenal syndrome).
  Urine samples take from patients via clean catch if the patient not have a catheter placed, otherwise take from urinary catheters if present. Straight catheterization utilize if the patient unable to void and doesn't have a catheter placed.
  Fecal specimens collect using a toilet specimen collection kit. Clinical, standart laboratory and cultural test, molecular genetic methods, using 16S rRNA gene sequencing of the V4-V5 hypervariable region be administered.
  Interventions: Diagnostic Test: 16S rRNA gene sequencing

INTERVENTIONS:
Diagnostic Test: 16S rRNA gene sequencing — DNA extraction and 16S rRNA gene sequencing DNA extraction, 16S rRNA gene amplification, and deep sequencing of the 16S rRNA amplicon performe.
  The V4-V5 region of the 16S rRNA gene amplify with barcodes for multiplexing.

SUMMARY:
Evaluate the prevalence and types of urinary tract infections, the features of the gut and urinary tract microbiota in cirrhosis, to assess its importance in the development of complications and outcomes of cirrhosis.

DETAILED DESCRIPTION:
Asymptomatic bacteriuria in an individual without urinary tract symptoms is defined by a mid-stream sample of urine showing bacterial growth > 105 cfu/mL in two consecutive samples in women and in one single sample in men. A complicated urinary tract infections occurs in an individual in whom factors related to the host (e.g. underlying diabetes or immunosuppression) or specific anatomical or functional abnormalities related to the urinary tract. Laboratory urine culture is the recommended method to determine the presence or absence of clinically significant bacteriuria.

Catheter-associated urinary tract infections refers to urinary tract infections occurring in a person whose urinary tract is currently catheterised or has been catheterised within the past 48 hours. Signs and systemic symptoms compatible with сatheter-associated urinary tract infections include new onset or worsening of fever, rigors, altered mental status, malaise, or lethargy with no other identified cause, flank pain, costovertebral angle tenderness, acute haematuria, pelvic discomfort and in those whose catheters have been removed dysuria, urgent or frequent urination and suprapubic pain or tenderness. Microbiologically, сatheter-associated urinary tract infections is defined by microbial growth of > 103 cfu/mL of one or more bacterial species in a single catheter urine specimen or in a mid-stream voided urine specimen from a patient whose urethral, suprapubic, or condom catheter has been removed within the previous 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cirrhosis

Exclusion Criteria:

* human immunodeficiency virus or acquired immune deficiency syndrome
* autoimmune diseases
* oncology
* organ transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational longitudinal multicenter study
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with variceal bleeding | from the date of assignment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 3 months
  The main diagnostic method of variceal bleeding is endoscopy
Number of Participants with hepatic coma | from the date of assignment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 3 months
  hepatic encephalopathy is graded with the West Haven Criteria: Grade 0 - No obvious changes other than a potentially mild decrease in intellectual ability and coordination Grade 1 - Trivial lack of awareness; euphoria or anxiety; shortened attention span; impaired performance of addition or subtraction Grade 2 - Lethargy or apathy; minimal disorientation for time or place; subtle personality change; inappropriate behaviour Grade 3 - Somnolence to semistupor, but responsive to verbal stimuli; confusion; gross disorientation Grade 4 - Coma
Number of Participants with hepatorenal syndrome | from the date of assignment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 3 months
  Type-1 hepatorenal syndrome is characterized by a rapid deterioration of renal function with a doubling of serum creatinine to values above 2.5 mg/dl within 2 weeks, type-2 hepatorenal syndrome is characterized by a slower increase in serum creatinine to values above 1.5 mg/dl. The main clinical characteristic of Type-1 hepatorenal syndrome is acute renal failure, while the main characteristic of type-2 hepatorenal syndrome is refractory ascites.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Stoma, D.Sc., Principal Investigator — Gomel State Medical University
Locations (1):
- Gomel State Clinical Hospital №3, Homyel, Ilicha Str. 286, Belarus

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) will no available to other researchers.

REFERENCES:
- [Result] Arvaniti V, D'Amico G, Fede G, Manousou P, Tsochatzis E, Pleguezuelo M, Burroughs AK. Infections in patients with cirrhosis increase mortality four-fold and should be used in determining prognosis. Gastroenterology. 2010 Oct;139(4):1246-56, 1256.e1-5. doi: 10.1053/j.gastro.2010.06.019. Epub 2010 Jun 14. PMID 20558165
- [Result] Mestrovic T, Matijasic M, Peric M, Cipcic Paljetak H, Baresic A, Verbanac D. The Role of Gut, Vaginal, and Urinary Microbiome in Urinary Tract Infections: From Bench to Bedside. Diagnostics (Basel). 2020 Dec 22;11(1):7. doi: 10.3390/diagnostics11010007. PMID 33375202
- [Result] Neugent ML, Hulyalkar NV, Nguyen VH, Zimmern PE, De Nisco NJ. Advances in Understanding the Human Urinary Microbiome and Its Potential Role in Urinary Tract Infection. mBio. 2020 Apr 28;11(2):e00218-20. doi: 10.1128/mBio.00218-20. PMID 32345639
- See also: In patients with cirrhosis, infections increase mortality 4-fold; 30% of patients die within 1 month after infection and another 30% die by 1 year. — https://pubmed.ncbi.nlm.nih.gov/20558165/
- See also: Consequently, studying the relationship between gut microbiota and the subsequent development of bacteriuria and UTI represents an important field of research. — https://pubmed.ncbi.nlm.nih.gov/33375202/
- See also: The contribution of the urinary tract microbiome to urinary tract infection and recurrent urinary tract infection — https://pubmed.ncbi.nlm.nih.gov/32345639/